CLINICAL TRIAL: NCT07291310
Title: Development of Cortical Plasticity Through Virtual Reality and Dual-Task Training in Children With Brachial Plexus Birth Injury: A Different Perspective in Paediatric Neurorehabilitation
Brief Title: Virtual Reality and Dual-Task Training for Cortical Plasticity in Children With Brachial Plexus Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Collaborators: Istanbul University (Other); Biruni University (Other)
Responsible Party: Principal Investigator, Barış CELBEK, Lecturer in Physiotherapy and Rehabilitation, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-BİAEK/14-49; 225S038 (Other Grant/Funding Number: TUBİTAK)
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Brachial Plexus Birth Palsy; Physical Therapy
Keywords: Brachial Plexus; Physiotherapy; Cortical Plasticity; Virtual Reality; Dual Task

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment design in which participants are randomly allocated to one of two intervention groups: a virtual reality-based exercise program or a dual-task motor-cognitive exercise program, both in addition to conventional physiotherapy
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Task Group (Experimental): Participants in the dual-task group will receive a motor-cognitive dual-task exercise program in addition to conventional physiotherapy. The program includes simultaneous motor activities (such as reaching, grasping, and upper-limb functional tasks) combined with cognitive challenges involving attention, memory, problem-solving, and decision-making. Each session lasts 60 minutes and is delivered three times per week for 12 weeks. The aim of the intervention is to enhance cortical activation, improve motor planning, and support upper-limb functional performance through combined motor and cognitive stimulation.
  Interventions: Other: Conventional Physiotherapy Program; Other: Dual Task
- Virtual reality (VR) Group (Experimental): Participants in the virtual reality (VR) group will receive a VR-based exercise program in addition to conventional physiotherapy. The VR program includes interactive upper-limb activities designed to promote active movement, motor control, and engagement through immersive, game-based tasks. Exercises target reaching, grasping, coordination, and proprioceptive awareness in a visually enriched environment. Each session lasts 60 minutes and is conducted three times per week for 12 weeks. The intervention aims to stimulate cortical activation, support motor learning, and enhance upper-limb functional performance.
  Interventions: Other: Conventional Physiotherapy Program; Other: Virtual Reality

INTERVENTIONS:
Other: Conventional Physiotherapy Program — The conventional physiotherapy program includes educating the child and family about the condition and treatment goals, maintaining regular communication, planning sessions according to the child's abilities, motivating the child, and promoting active participation. Exercises are designed based on functional, daily-life, and play activities to maintain attention and engagement, following El-Shamy et al. (2017).
  Before each session, a 15-minute warm-up of shoulder internal rotation, pectoral, and elbow extension stretches will be performed (3 sets of 10 repetitions, 5-second hold).
Other: Virtual Reality — Children in the VR group will perform conventional physiotherapy followed by 20 minutes of VR-based exercises using the Becure Leap Motion system. The games involve interactive tasks designed to improve wrist, hand, and upper-limb movements, coordination, and motor control, with progressively increasing difficulty levels. Sessions are supervised by the study physiotherapist.
  Arms: Virtual reality (VR) Group
Other: Dual Task — Children in the dual-task group will perform exercises integrating conventional physiotherapy with cognitive-motor dual-task activities for a total of 45 minutes per session, following Wollesen et al. (2022). Cognitive tasks will be age- and ability-appropriate: younger children will perform basic memory and attention tasks, while older children will engage in more complex problem-solving, rapid decision-making, and language-based tasks.
  Task selection will consider the impact on motor performance, including movement quality, divided attention, reaction time, coordination, and executive functions, aiming to maximize motor-cognitive interaction. To maintain motivation, tasks will be gamified, competitive, offer choices based on personal interest, provide feedback, and reward achievements. Task difficulty will be adjusted individually.
  Arms: Dual Task Group

SUMMARY:
Brachial plexus birth injury (BPBI) is a condition that occurs when the nerves controlling the arm are injured during birth, leading to weakness, limited movement, and sensory problems. These motor difficulties may also affect cognitive processes related to movement. BPBI requires long-term follow-up and rehabilitation.

This study will compare two treatment approaches in children with BPBI:

* virtual reality (VR)-based exercises, and
* motor-cognitive dual-task exercises. We will examine their effects on brain adaptation (cortical activation), muscle strength, joint motion, proprioception, and upper-limb function. Fourteen children aged 7-14 years will be randomly assigned to one of the two programs, each delivered for 12 weeks. Afterward, participants will continue a 9-month home program. Assessments will be conducted at baseline, after treatment, and at 12 months, including functional MRI (fMRI).

This study will be the first to evaluate long-term brain changes and functional outcomes after these two rehabilitation approaches in children with BPBI.

DETAILED DESCRIPTION:
Brachial plexus birth injury (BPBI) is characterized by unilateral or bilateral upper extremity motor and sensory impairment resulting from injury to the cervical (C4-C5 to T1-T2) nerve roots and their associated structures during birth. BPBI often leads to limited active movement, muscle weakness, impaired proprioception, and secondary musculoskeletal problems. Beyond these peripheral symptoms, decreased use of the affected limb and chronic motor impairment may influence cognitive processes related to motor planning and execution. Recent literature also highlights the role of central nervous system plasticity in functional recovery; however, evidence remains limited, and long-term cortical adaptation patterns in children with BPBI are not well understood.

This randomized controlled study aims to compare the effects of two rehabilitation approaches-virtual reality (VR)-based exercises and motor-cognitive dual-task exercises-on cortical adaptation, joint range of motion, muscle strength, proprioception, and upper extremity function in children with BPBI. A secondary aim is to examine the relationship between cortical activation and functional performance.

A total of 14 children aged 7-14 years with C5-C6 or C5-C7 involvement, who have not undergone neurosurgery and score ≥26 on the Modified Pediatric Mini Mental Scale, will be included. Participants will be randomly allocated into two groups:

1. VR-based exercise + conventional physiotherapy (n = 7),
2. Dual-task motor-cognitive exercise + conventional physiotherapy (n = 7).

Interventions will be delivered for 12 weeks, three sessions per week, with each session lasting 1 hour. After the supervised intervention period, participants will continue with a structured home program for 9 months. Evaluations will be conducted at baseline, post-intervention (12 weeks), and at 12 months. Cortical activation will be assessed using functional magnetic resonance imaging (fMRI). Additional outcome measures will include joint range of motion, muscle strength, proprioception, Modified Mallet Classification, and the Brachial Plexus Outcome Measure.

This study is designed to provide novel insights into neuroplastic changes associated with two different rehabilitation approaches and to clarify long-term associations between cortical activation and functional recovery. The findings are expected to contribute to the development of multidisciplinary, neuromodulatory rehabilitation strategies aimed at improving upper extremity function and overall quality of life in children with BPBI.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-14 years
* Diagnosed with unilateral DBPP
* C5-C6 or C5-C7 involvement (Narakas I, IIa, IIb)
* Modified Pediatric Mini-Mental Scale score ≥26
* Child and parent willing to participate in the study

Exclusion Criteria:

* Previous nerve surgery for DBPP
* Surgery within the past year or Botulinum Toxin injection within the past 3 months
* Any neurological condition other than DBPP
* Vision or hearing impairments affecting participation
* Contraindications for fMRI
* Fixed contractures in shoulder, elbow, wrist, or finger joints
* Participation in regular physiotherapy or other rehabilitation programs within the past 3 months

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Motor Cortex Activation (BOLD Signal) Measured by fMRI | From baseline (pre-treatment) to 12 weeks of intervention and 9-month follow-up after baseline.
  Motor cortex activation will be evaluated before treatment, after 12 weeks, and at 9-month follow-up using non-contrast BOLD fMRI during finger and elbow movements to assess cortical plasticity.
Range of Motion (ROM) | From baseline (pre-treatment) to 12 weeks of intervention and 9 months follow-up after baseline.
  Active joint movement of the affected upper limb will be measured with an electronic goniometer in standardized positions for shoulder, elbow, and wrist.
Brachial Plexus Outcome Measure (BPOM) | From baseline (pre-treatment) to 12 weeks of intervention and 9 months follow-up after baseline.
  Functional performance of the upper limb in daily activities will be assessed using a validated scale, including shoulder, elbow, and hand tasks. The BPOM consists of three domains (shoulder, elbow, and hand) and includes 11 task-based activities, each scored on a 5-point scale (1-5). The total BPOM score ranges from 11 to 55, with higher scores indicating better upper limb functional performance.
Muscle Strength | From baseline (pre-treatment) to 12 weeks of intervention and 9 months follow-up after baseline.
  Upper limb muscle groups will be tested using a handheld dynamometer with standardized positions and the "make method."

SECONDARY OUTCOMES:
Change in Joint Position Sense Error (Degrees) of the Upper Limb Measured | From baseline (pre-treatment) to 12 weeks of intervention and 9 months follow-up after baseline.
  Joint position sense for shoulder, elbow, and wrist will be evaluated using a KForce Sens® device, comparing target and replicated angles with eyes closed.
Modified Mallet Classification | From baseline (pre-treatment) to 12 weeks of intervention and 9 months follow-up after baseline
  Global upper limb movement patterns and functional ability will be assessed using 5 key shoulder and hand tasks, scored 1-5.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Hoşbay, Principal Investigator — Biruni University

IPD SHARING:
Plan to Share IPD: No